CLINICAL TRIAL: NCT05289791
Title: The Effect of Ultrasonic Activation of Bioceramic Sealer on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Effect of Ultrasonic Activation of Bioceramic Sealer on Postoperative Pain in Lower Premolars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant Yasser Shaker Ibrahim El-Saharty, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-3-5
Record Dates: First submitted 2022-03-09; First posted 2022-03-21 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasonic activation of bioceramic sealer (Experimental): ultrasonic activation of bioceramic sealer for 20 seconds
  Interventions: Other: ultrasonic activation of bioceramic sealer
- bioceramic sealer (Active Comparator): bioceramic sealer
  Interventions: Other: ultrasonic activation of bioceramic sealer

INTERVENTIONS:
Other: ultrasonic activation of bioceramic sealer — activation of bioceramic sealer using ultrasonic tip for 20 seconds in buccolingual and mesiodistal direction

SUMMARY:
The aim of this study is to clinically compare post-operative pain levels after ultrasonic activation of Ceraseal bioceramic sealer versus non-activated bioceramic sealer for patients with symptomatic irreversible pulpitis related to mandibular premolar teeth.

DETAILED DESCRIPTION:
To clinically compare post-operative pain levels after ultrasonic activation of Ceraseal bioceramic sealer versus non-activated bioceramic sealer for patients with symptomatic irreversible pulpitis related to mandibular premolar teeth.Ultrasonic activation of Ceraseal bioceramic sealer for 20 seconds using non cutting ultrasonic tip.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old and to 50.
* Male or female.
* Patients seeking root canal treatment.
* Mandibular posterior teeth with Symptomatic irreversible pulpitis with preoperative sharp, moderate, or severe pain with normal periapical radiographic appearance or slight widening in lamina dura.
* Systematically healthy patient (ASA I, II).
* Patient who can understand modified VAS and sign informed consent

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders. (ASA III or IV).
* History of intolerance to NSAIDS.
* Patients with two or more adjacent teeth requiring endodontic treatment.
* External root resorption.
* Internal root resorption.
* Vertical root fracture.
* Periapical lesion.
* Association with swelling.
* Acute peri-apical abscess or acute exacerbation of a chronic abscess.
* Pregnancy.
* Use of ibuprofen in the last 12 hour.
* Bleeding disorder.
* Long term corticosteroid use.
* Mobility Grade II or III.
* Pocket depth more than 5mm.
* Previous root canal therapy.
* Non-restorability.
* TMJ problems, bruxism, clenching or traumatic occlusion.
* Inability to perceive the given instructions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 6 hours
  intensity of pain on modified Visual analogue scale
postoperative pain | 12 hours
  intensity of pain on modified Visual analogue scale
postoperative pain | 24 hours
  intensity of pain on modified Visual analogue scale
postoperative pain | 48 hours
  intensity of pain on modified Visual analogue scale

SECONDARY OUTCOMES:
number of analgesic tablets taken by patient after endodontic treatment | up to 48 hours postoperatively
  number of analgesics taken by patient in 1st 48 hours
Sealer Extrusion laterally and periapically | Immediately after obturation.
  presence or absence of sealer extrusion

CONTACTS AND LOCATIONS:
Overall Officials: Heba M. El-far, professor, Study Director — Cairo University
Locations (1):
- Cairo university, Giza, Manial, Egypt